CLINICAL TRIAL: NCT00999609
Title: A Safety and Efficacy Study in Subjects With Leber Congenital Amaurosis (LCA) Using Adeno-Associated Viral Vector to Deliver the Gene for Human RPE65 to the Retinal Pigment Epithelium (RPE) [AAV2-hRPE65v2-301]
Brief Title: Safety and Efficacy Study in Subjects With Leber Congenital Amaurosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Collaborators: Children's Hospital of Philadelphia (Other); University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAV2-hRPE65v2-301
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Inherited Retinal Dystrophy Due to RPE65 Mutations; Leber Congenital Amaurosis
Keywords: Adeno-associated virus; AAV; Leber congenital amaurosis; RPE65; Gene therapy; Gene transfer; voretigene neparvovec-rzyl; Retinitis pigmentosa
MeSH Terms: conditions — Leber Congenital Amaurosis; Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AAV2-hRPE65v2,voretigene neparvovec-rzyl (Experimental): voretigene neparvovec rzyl, 1.5 E11 vector genomes, per eye, administered by subretinal injection in a volume of 0.3mL, 6-18 days apart
  Interventions: Biological: AAV2-hRPE65v2,voretigene neparvovec-rzyl
- Control (No Intervention): No intervention

INTERVENTIONS:
Biological: AAV2-hRPE65v2,voretigene neparvovec-rzyl — Subretinal administration of gene therapy vector AAV2-hRPE65v2 (1.5E11 vector genomes per eye) to both eyes via surgical procedures on separate days.
  Other Names: AAV2-hRPE65v2; voretigene neparvovec-rzyl; gene therapy vector
  Arms: AAV2-hRPE65v2,voretigene neparvovec-rzyl

SUMMARY:
The study is a Phase 3, open-label, randomized controlled trial of gene therapy intervention by subretinal administration of AAV2-hRPE65v2 (voretigene neparvovec-rzyl). At least twenty-four subjects, three years of age or older, will be recruited. The intervention group will receive AAV2-hRPE65v2 at either The Children's Hospital of Philadelphia or University of Iowa to determine if it improves visual and retinal function in individuals with RPE65 gene mutations.

DETAILED DESCRIPTION:
Leber congenital amaurosis (LCA) is a disease where part of the eye (the retina) is severely diseased. Usually it is detected in affected people within the first few months of life, as there is significantly poor vision at birth. Cells in the retina are lost over time in people with LCA, which typically leads to total blindness. There are no pharmacological treatments available. This study will focus on the form of LCA caused by changes (mutations) in DNA that makes a certain protein (called the 65 kDa retinal pigment epithelium (RPE)-specific protein, or RPE65). This can be confirmed by a special method of testing (molecular testing) to verify the presence of RPE65 gene mutations.

This study uses a gene therapy vector made from an adeno-associated virus (AAV) called AAV2-hRPE65v2 (voretigene neparovec-rzyl). Gene therapy refers to the incorporation of new DNA into cells with the goal of supplying a therapeutic gene or a gene that is missing or not functioning in the cell. The AAV parts of the gene therapy vector work as a delivery vehicle for providing the normal human RPE65 gene to the cells of the retina. An earlier Phase 1 clinical study of AAV2-hRPE65v2 was conducted based on the demonstration of safety and effectiveness of the vector in animals with a similar eye disease. The earlier Phase 1 clinical study was a dose-escalation study primarily designed to evaluate safety in humans, and tested three doses of the vector in twelve children and adults. The safety of injecting into the second eye was also evaluated. The results from these earlier Phase 1 studies showed an acceptable safety profile.

This study will deliver AAV2-hRPE65v2 vector (voretigene neparvovec-rzyl) to at least sixteen intervention group subjects, age three or older; subjects will receive the vector in both eyes via subretinal injections during surgeries (on separate days). The purpose of this research study is to assess the efficacy and safety of the AAV2-hRPE65v2 gene therapy vector (voretigene neparvovec-rzyl) as a possible treatment for LCA due to RPE65 gene mutations. The control group of at least eight subjects will be able to cross-over to the intervention group after one year, provided they still meet all eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to adhere to protocol and long-term follow-up as evidenced by written informed consent or parental permission and subject assent (where applicable).
* Diagnosis of LCA due to RPE65 mutations; molecular diagnosis is to be performed, or confirmed, by a CLIA-approved laboratory.
* Age three years old or older.
* Visual acuity worse than 20/60 (both eyes) and/or visual field less than 20 degrees in any meridian as measured by a III4e isopter or equivalent (both eyes).
* Sufficient viable retinal cells as determined by non-invasive means, such as optical coherence tomography (OCT) and/or ophthalmoscopy. Must have either: 1) an area of retina within the posterior pole of >100 µm thickness shown on OCT; 2) ≥ 3 disc areas of retina without atrophy or pigmentary degeneration within the posterior pole; or 3) remaining visual field within 30 degrees of fixation as measured by a III4e isopter or equivalent.
* Subjects must be evaluable on mobility testing (the primary efficacy endpoint) to be eligible for the study. Evaluable is defined as: 1) The ability to perform mobility testing within the luminance range evaluated in the study. Individuals must receive an accuracy score of ≤ 1 during screening mobility testing at 400 lux or less to be eligible; individuals with an accuracy score of > 1 on all screening mobility test runs at 400 lux, or those who refuse to perform mobility testing at screening, will be excluded. 2) The inability to pass mobility testing at 1 lux. Individuals must fail screening mobility testing at 1 lux to be eligible; individuals that pass one or more screening mobility test runs at 1 lux will be excluded.

Exclusion Criteria:

* Unable or unwilling to meet requirements of the study, including receiving bilateral subretinal vector administrations.
* Any prior participation in a study in which a gene therapy vector was administered.
* Participation in a clinical study with an investigational drug in the past six months.
* Use of retinoid compounds or precursors that could potentially interact with the biochemical activity of the RPE65 enzyme; individuals who discontinue use of these compounds for 18 months may become eligible.
* Prior intraocular surgery within six months.
* Known sensitivity to medications planned for use in the peri-operative period.
* Pre-existing eye conditions or complicating systemic diseases that would preclude the planned surgery or interfere with the interpretation of study. Complicating systemic diseases would include those in which the disease itself, or the treatment for the disease, can alter ocular function. Examples are malignancies whose treatment could affect central nervous system function (for example: radiation treatment of the orbit; leukemia with CNS/optic nerve involvement). Subjects with diabetes or sickle cell disease would be excluded if they had any manifestation of advanced retinopathy (e.g., macular edema or proliferative changes). Also excluded would be subjects with immunodeficiency (acquired or congenital) as there could be susceptibility to opportunistic infection (such as CMV retinitis).
* Individuals of childbearing potential who are pregnant or unwilling to use effective contraception for four months following vector administration.
* Individuals incapable of performing mobility testing (the primary efficacy endpoint) for reason other than poor vision, including physical or attentional limitations.
* Any other condition that would not allow the potential subject to complete follow-up examinations during the course of the study or, in the opinion of the investigator, makes the potential subject unsuitable for the study.
* Subjects will not be excluded based on their gender, race, or ethnicity.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2030-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Albert M Maguire, MD, Principal Investigator — Children's Hospital of Philadelphia; Stephen R Russell, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Maguire AM, Simonelli F, Pierce EA, Pugh EN Jr, Mingozzi F, Bennicelli J, Banfi S, Marshall KA, Testa F, Surace EM, Rossi S, Lyubarsky A, Arruda VR, Konkle B, Stone E, Sun J, Jacobs J, Dell'Osso L, Hertle R, Ma JX, Redmond TM, Zhu X, Hauck B, Zelenaia O, Shindler KS, Maguire MG, Wright JF, Volpe NJ, McDonnell JW, Auricchio A, High KA, Bennett J. Safety and efficacy of gene transfer for Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2240-8. doi: 10.1056/NEJMoa0802315. Epub 2008 Apr 27. PMID 18441370
- [Background] Maguire AM, High KA, Auricchio A, Wright JF, Pierce EA, Testa F, Mingozzi F, Bennicelli JL, Ying GS, Rossi S, Fulton A, Marshall KA, Banfi S, Chung DC, Morgan JI, Hauck B, Zelenaia O, Zhu X, Raffini L, Coppieters F, De Baere E, Shindler KS, Volpe NJ, Surace EM, Acerra C, Lyubarsky A, Redmond TM, Stone E, Sun J, McDonnell JW, Leroy BP, Simonelli F, Bennett J. Age-dependent effects of RPE65 gene therapy for Leber's congenital amaurosis: a phase 1 dose-escalation trial. Lancet. 2009 Nov 7;374(9701):1597-605. doi: 10.1016/S0140-6736(09)61836-5. Epub 2009 Oct 23. PMID 19854499
- [Background] Chung DC, McCague S, Yu ZF, Thill S, DiStefano-Pappas J, Bennett J, Cross D, Marshall K, Wellman J, High KA. Novel mobility test to assess functional vision in patients with inherited retinal dystrophies. Clin Exp Ophthalmol. 2018 Apr;46(3):247-259. doi: 10.1111/ceo.13022. Epub 2017 Aug 31. PMID 28697537
- [Background] Chung DC, Bertelsen M, Lorenz B, Pennesi ME, Leroy BP, Hamel CP, Pierce E, Sallum J, Larsen M, Stieger K, Preising M, Weleber R, Yang P, Place E, Liu E, Schaefer G, DiStefano-Pappas J, Elci OU, McCague S, Wellman JA, High KA, Reape KZ. The Natural History of Inherited Retinal Dystrophy Due to Biallelic Mutations in the RPE65 Gene. Am J Ophthalmol. 2019 Mar;199:58-70. doi: 10.1016/j.ajo.2018.09.024. Epub 2018 Sep 28. PMID 30268864
- [Result] Ashtari M, Cyckowski LL, Monroe JF, Marshall KA, Chung DC, Auricchio A, Simonelli F, Leroy BP, Maguire AM, Shindler KS, Bennett J. The human visual cortex responds to gene therapy-mediated recovery of retinal function. J Clin Invest. 2011 Jun;121(6):2160-8. doi: 10.1172/JCI57377. Epub 2011 May 23. PMID 21606598
- [Result] Simonelli F, Maguire AM, Testa F, Pierce EA, Mingozzi F, Bennicelli JL, Rossi S, Marshall K, Banfi S, Surace EM, Sun J, Redmond TM, Zhu X, Shindler KS, Ying GS, Ziviello C, Acerra C, Wright JF, McDonnell JW, High KA, Bennett J, Auricchio A. Gene therapy for Leber's congenital amaurosis is safe and effective through 1.5 years after vector administration. Mol Ther. 2010 Mar;18(3):643-50. doi: 10.1038/mt.2009.277. Epub 2009 Dec 1. PMID 19953081
- [Result] Bennett J, Ashtari M, Wellman J, Marshall KA, Cyckowski LL, Chung DC, McCague S, Pierce EA, Chen Y, Bennicelli JL, Zhu X, Ying GS, Sun J, Wright JF, Auricchio A, Simonelli F, Shindler KS, Mingozzi F, High KA, Maguire AM. AAV2 gene therapy readministration in three adults with congenital blindness. Sci Transl Med. 2012 Feb 8;4(120):120ra15. doi: 10.1126/scitranslmed.3002865. PMID 22323828
- [Result] Russell S, Bennett J, Wellman JA, Chung DC, Yu ZF, Tillman A, Wittes J, Pappas J, Elci O, McCague S, Cross D, Marshall KA, Walshire J, Kehoe TL, Reichert H, Davis M, Raffini L, George LA, Hudson FP, Dingfield L, Zhu X, Haller JA, Sohn EH, Mahajan VB, Pfeifer W, Weckmann M, Johnson C, Gewaily D, Drack A, Stone E, Wachtel K, Simonelli F, Leroy BP, Wright JF, High KA, Maguire AM. Efficacy and safety of voretigene neparvovec (AAV2-hRPE65v2) in patients with RPE65-mediated inherited retinal dystrophy: a randomised, controlled, open-label, phase 3 trial. Lancet. 2017 Aug 26;390(10097):849-860. doi: 10.1016/S0140-6736(17)31868-8. Epub 2017 Jul 14. PMID 28712537
- [Derived] Fischer MD, Simonelli F, Sahni J, Holz FG, Maier R, Fasser C, Suhner A, Stiehl DP, Chen B, Audo I, Leroy BP; PERCEIVE Study Group. Real-World Safety and Effectiveness of Voretigene Neparvovec: Results up to 2 Years from the Prospective, Registry-Based PERCEIVE Study. Biomolecules. 2024 Jan 17;14(1):122. doi: 10.3390/biom14010122. PMID 38254722
- [Derived] Bhadhuri A, Droschel D, Guldimann M, Jetschgo C, Banhazi J, Schwenkglenks M, Sutherland CS. Cost-effectiveness of voretigene neparvovec in the treatment of patients with inherited retinal disease with RPE65 mutation in Switzerland. BMC Health Serv Res. 2022 Jun 28;22(1):837. doi: 10.1186/s12913-022-08211-y. PMID 35765055

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Bilateral subretinal injection of voretigene neparvovec-rzyl (AAV2-hRPE65v2), 1.5x 10e11 vg in a total volume of 0.3ml per eye, administered no fewer than 6 days apart
- Control: No intervention, no sham; uninjected control group
Period: Overall Study
Arm/Group | Intervention | Control
Started | 21 (Before intervention) | 10
Completed | 20 (1 year post intervention) | 9 (1 year post intervention)
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control: Control group did not receive voretigene neparvovec-rzyl. The control group became eligible to receive voretigene neparvovec-rzyl 1 year after their baseline evaluations, provided they still met all eligibility criteria.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (11.8) | 15.9 (9.5) | 15.1 (10.9)
Age, Customized [Count of Participants; unit: Participants]
  Age Group: <10 years old | 9 | 4 | 13
  Age Group: ≥10 years old | 12 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 16 | 9 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 7 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Multi-luminance Mobility Test (MLMT), bilateral, passing at a lux level of < 125 or ≥ 125 lux [Count of Participants; unit: Participants] — The multi-luminance mobility test (MLMT) measures changes in functional vision, based on the ability to navigate a course accurately and at a reasonable pace at different levels of environmental illumination. The MLMT was assessed at 1 or more of 7 light levels ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night). At baseline, stratification was based on the lowest passing light level (less than or equal to 125 lux or greater than 125 lux).
  Participants
    Lowest passing light level of < 125 lux | 12 | 4 | 16
    Lowest passing light level of ≥ 125 lux | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Multi-luminance Mobility Testing (MLMT), Bilateral
Description: The MLMT measures changes in functional vision, as assessed by the ability to navigate a course accurately and at a reasonable pace at different levels of environmental illumination. MLMT was assessed using both eyes at 1 or more of 7 levels of illumination, ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night). Each light level was assigned a score code ranging from 0 to 6. A higher score indicated that a subject was able to pass the MLMT at a lower light level. A score of -1 was assigned to those who could not pass MLMT at 400 lux. The MLMT of each subject was videotaped and assessed by independent graders. The MLMT score was determined by the lowest light level at which the subject was able to pass the MLMT. The MLMT score change was defined as the difference between the score at Baseline and the score at Year 1. A positive MLMT score change from Baseline to Year 1 visit indicated that the subject was able to complete the MLMT at a lower light level.
Time Frame: One year (change from baseline)
Measure: Mean (Standard Deviation); unit: Score Change in Light Levels
Groups:
- Intervention: Bilateral, subretinal injection of voretigene neparvovec-rzyl (AAV2-hRPE65v2)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 10
Score Change in Light Levels | 1.8 (1.1) | 0.2 (1.0)

2. Secondary Outcome: Full-field Light Sensitivity Threshold (FST) Testing: White Light
Description: Measures the light sensitivity of the entire visual field by recording the luminance at which a subject reliably reports seeing the dimmest flash.
Time Frame: One year (change from baseline)
Measure: Mean (Standard Error); unit: log10(cd.s/(m^2))
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 10
log10(cd.s/(m^2)) | -2.08 (0.29) | 0.04 (0.44)

3. Secondary Outcome: Multi-luminance Mobility Testing (Monocular)
Description: The MLMT measures changes in functional vision, as assessed by the ability to navigate a course accurately and at a reasonable pace at different levels of environmental illumination. MLMT was assessed using the first eye at 1 or more of 7 levels of illumination, ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night). Each light level was assigned a score code ranging from 0 to 6. A higher score indicated that a subject was able to pass the MLMT at a lower light level. A score of -1 was assigned to those who could not pass MLMT at 400 lux. The MLMT of each subject was videotaped and assessed by independent graders. The MLMT score was determined by the lowest light level at which the subject was able to pass the MLMT. The MLMT score change was defined as the difference between the score at Baseline and the score at Year 1. A positive MLMT score change from Baseline to Year 1 visit indicated that the subject was able to complete the MLMT at a lower light level.
Time Frame: One year (change from baseline)
Measure: Mean (Standard Deviation); unit: Score Change in Light Levels
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 10
Score Change in Light Levels | 1.9 (1.2) | 0.2 (0.6)

4. Secondary Outcome: Visual Acuity
Description: Measurement of the sharpness of vision, determined by the ability to read letters on a standardized chart from a specified distance.
Time Frame: One year (change from baseline)
Measure: Mean (Standard Error); unit: LogMAR
Arm/Group | Intervention | Control
Number analyzed (Participants) | 21 | 10
LogMAR | -0.16 (0.07) | 0.01 (0.10)

ADVERSE EVENTS:
Time Frame: 1 year post administration (Intervention group), 1 year post baseline (Control group)
Description: The safety population (n=29) includes all subjects who received injection in either eye for the intervention group and all control group subjects who did not withdraw, or were not withdrawn, prior to any of the following people knowing the treatment assignment: the subject, parent, Principal Investigator, or Medical Monitor.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/9
Other Adverse Events (participants affected / at risk) | 13/20 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=20) | Control (N=9)
Adverse Drug Reaction (Surgical and medical procedures) | 2 (2) | 0 (0) — Associated with pre-existing complex seizure disorder and complications of oral surgery, respectively
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) — Associated with pre-existing complex seizure disorder.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=20) | Control (N=9)
Cataract (Eye disorders) | 3 (4) | 0 (0)
Elevated intraocular pressure (Eye disorders) | 4 (5) | 0 (0)
Retinal tear (Eye disorders) | 2 (2) | 0 (0)
Eye inflammation (Eye disorders) | 2 (6) | 0 (0)
Conjunctival cyst (Eye disorders) | 1 (1) | 0 (0)
Conjunctivis viral (Eye disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Macular hole/degeneration (Eye disorders) | 1 (2) | 0 (0) — Same eye of a single subjects, a full-thickness macular hole spontaneously resolved (with sequelae) to thinning, which subsequently resolved (without sequelae). Classified as two adverse events, but occurred in the same clinical course of events.
Maculopathy/ epiretinal membrane (Eye disorders) | 1 (2) | 0 (0)
Pseudopapilledema (Eye disorders) | 1 (1) | 0 (0)
Retinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes